CLINICAL TRIAL: NCT03870633
Title: Assessing Financial Difficulty in Patients with Blood Cancers
Brief Title: Assessment of Financial Difficulty in Participants with Chronic Lymphocytic Leukemia and Multiple Myeloma
Status: Completed | Type: Observational
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH); The Leukemia and Lymphoma Society (Other)
Responsible Party: Sponsor
Other Study IDs: A231602CD; NCI-2018-01708 (Registry Identifier: NCI Clinical Trial Reporting Program); UG1CA189823 (NIH)
Record Dates: First submitted 2019-02-26; First posted 2019-03-12 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Chronic Lymphocytic Leukemia; Plasma Cell Myeloma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Multiple Myeloma | interventions — Interviews as Topic; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational (medical chart, interview): Participants undergo medical chart abstraction within 1 week and complete telephone interview over 30-45 minutes within 8 weeks after registration.
  Interventions: Other: Medical Chart Review; Other: Interview; Other: Questionnaire; Other: Quality-of-Life Assessment

INTERVENTIONS:
Other: Medical Chart Review — Undergo medical chart abstraction
Other: Interview — Complete telephone interview
Other: Questionnaire — Ancillary studies
Other: Quality-of-Life Assessment — Ancillary studies

SUMMARY:
This trial studies financial difficulty in participants with chronic lymphocytic leukemia and multiple myeloma. Assessment of financial difficulty may help to better understand the financial impact of cancer and come up with ways to help participants avoid financial problems during treatment.

DETAILED DESCRIPTION:
The primary and secondary objectives of the study:

PRIMARY OBJECTIVES:

I. To estimate the proportion of patients with multiple myeloma (MM) or chronic lymphocytic leukemia (CLL) who report experiencing financial difficulty in the past 12 months.

SECONDARY OBJECTIVES:

I. To describe the association of patient report of financial difficulty with insurance status.

II. To describe the association of patient report of financial difficulty with receiving treatment at sites of care that report offering patients financial guidance through navigators or social workers, and controlling for patient socioeconomic status.

III. To describe the types of psychosocial, transportation and financial navigation interventions sites are developing.

IV. To identify distinct patterns of financial burden among patients undergoing treatment for MM or CLL.

V. To examine the relationship between distinct patterns of financial burden with patient report of financial difficulty, patient socio-demographics, and patient disease characteristics.

VI. To estimate the proportion of patients with MM or CLL undergoing treatment who report receiving financial support in the past 12 months.

VII. To describe the association of patient report of receiving financial support with receiving treatment at sites of care offering patients financial guidance through navigators or social workers, and with socioeconomic status.

VIII. To describe the magnitude of patient concerns regarding treatment and costs of care.

IX. To describe the association of patient concerns regarding treatment and costs of care with patient socio-demographics, disease and site of care characteristics.

X. To describe the association of financial difficulty with patient self-reported health and well-being.

Trial Design:

OUTLINE:

Participants undergo medical chart abstraction within 1 week and complete telephone interview over 30-45 minutes within 8 weeks after registration.

ELIGIBILITY:
Inclusion Criteria:

PATIENT ELIGIBILITY CRITERIA

* Patients must have current diagnosis of chronic lymphocytic leukemia (CLL) or multiple myeloma (MM)
* Patients' medical records must be available to the registering institution
* Eligible patients must have been prescribed drug-based anticancer therapy, whether administered orally or by infusion, within the prior 12 months. Specifically, eligible patients are those who:

  * Are presently being treated with infused or orally-administered anticancer therapy, OR
  * Completed infused or orally-administered anti-cancer therapy in the past 12 months, OR
  * Were prescribed infused or orally-administered anticancer therapy within the prior 12 months yet chose to forego treatment
* Not currently enrolled in a clinical trial in which drug is supplied by the study
* Patients with psychiatric illness or other mental impairment that would preclude their ability to give informed consent or to respond to the telephone survey are not eligible
* Patients must be able to read and comprehend English or Spanish

SITE ELIGIBILITY CRITERIA

* Intent to complete the A231602CD Site of Care Survey
* Access to patient medical records: Registering institution must have access to patient medical records, either on site or via request from other institutions, if recruiting patients at a site (as medical abstraction is required for collecting study data)
* Sites seeking to enroll Spanish- speaking patients must have Spanish speaking staff on site to be able to conduct the informed consent discussion in Spanish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with a current diagnosis of CLL or MM with medical records available to the registering institution
Sampling Method: Non-Probability Sample
Enrollment: 521 (Actual)
Dates: Start 2019-05-14 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with MM and/or CLL who report experiencing financial difficulties in the past 12 months | Up to 8 weeks
  Financial difficulties will be assessed using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) financial difficulty item #28 regarding financial difficulties with a modified recall period: "Has your physical condition or medical treatment caused you financial difficulties in the past year?", measured as "Not at all/A little/Quite a bit/Very much." Participant responses will be dichotomized as follows: "Not at all" or "A little" classified as "No", and "Quite a bit" and "very much" classified as "Yes." This dichotomized response will be assessed using Wilson score confidence interval (95%).

SECONDARY OUTCOMES:
Association of insurance status with financial difficulties in the past 12 months assessed with the EORTC QLQ-C30 financial difficulty item | Up to 8 weeks
  The association of patient report of financial difficulty as measured by the EORTC QLQ-C30 item #28 regarding financial difficulties with a modified recall period: "Has your physical condition or medical treatment caused you financial difficulties in the past year?" with insurance status (defined as those with Medicare/Medicaid v. those with commercial insurance) will be assessed using Mann-Whitney U test. Item #28 on the EORTC QLQ-C30 is measured as "Not at all/A little/Quite a bit/Very much", converted to 0, 1, 2 and 3 respectively for the purposes of analysis.
Association of financial difficulties in the past 12 months assessed with the EORTC QLQ-C30 and receiving treatment at practices that report offering patients financial guidance. | Up to 8 weeks
  The association of patient report of financial difficulty as measured by the EORTC QLQ-C30 item #28 with receiving treatment at sites of care that report offering patients financial guidance through navigators or social workers as measured by question 20 of the protocol practice survey will be tested using multinomial logistic regression modeling. In this model the outcome will be the patient report of financial difficulty, and the covariates will be the financial guidance questions from the protocol practice survey, along with disease/treatment characteristics and indicators of patient socioeconomic status. Question 20 of the protocol practice survey asks the site to state the financial navigation services that are currently offered at their practice to all cancer patients or their families. If a site offers at least one service, they will be treated as offering financial guidance (measured as "Yes/No").
Association of financial difficulties in the past 12 months assessed with the EORTC QLQ-C30 and patient socioeconomic status | Up to 8 weeks
  The association of patient socioeconomic status (as measured by part 3, question 6 of the patient protocol survey) and patient reported financial difficulty (as measured by item #28 of the EORTC QLQ-C30) will be tested using multinomial logistic regression modeling. In this model the outcome will be the patient report of financial difficulty, and the covariates will be the patient reported total household income. Item #28 on the EORTC QLQ-C30 is measured as "Not at all/A little/Quite a bit/Very much", converted to 0, 1, 2 and 3 respectively for the purposes of analysis. Part 3, question 6 of the patient protocol survey asks the patient to state the total income of the household they live in and is measured with the following options: less than $20,000, $20,000 - 39,999, $40,000 - 59,999, $60,000 - 79,999, $80,000 - 99,999, $100,000 or more, Don't know.
Financial support evaluated using site-reported plans of developing psychosocial, transportation and financial navigation services found in the Site of Care Survey | Up to 8 weeks
  Descriptive statistics will be used to describe the site-reported plans of developing psychosocial (question 46 of the protocol site survey), transportation (question 33 of the protocol site survey), and financial navigation services (question 24 of the protocol site survey). Each of these questions asks the site to state if they have plans to develop or enhance psychosocial, transportation or financial navigation services (all answered as "Yes/No" questions).
Identify distinct patterns of financial burden assessed with the EORTC QLQ-C30 among patients undergoing treatment for MM and/or CLL | Up to 8 weeks
  Patterns of financial difficulty (item #28 of the EORTC QLQ-C30) will be assessed utilizing measures of patient reported difficulties paying medical bills (part 1, question 1), delays or foregoing treatment (as measured by part 1, question 4), difficulties covering non-medical expenses due to costs of treatment (part 1, question 7), and financial worries (part 1,). Exploratory LCA will be conducted to assess these patterns. Question 1 asks the participant if they had any problems paying any medical bills in the last twelve months (Yes/No). Question 4 asks the participant if they y delayed medical care because they were worried about the cost (Yes/No). Question 7asks the participant if they had to make any sacrifices in the past 5 years because of debt related to medical care (Yes/No). Question 9 asks the participant if they get sicker or have an accident, how worried are they that they will not be able to pay for their medical bills (Very, Somewhat or Not worried).
To examine the relationship between distinct patterns of patient-reported financial burden with patient report of financial difficulty, with patient socio-demographics, and with patient disease characteristics. | Up to 8 weeks
  This analysis will identify the relationship between distinct patterns of financial burden (as measured by part 1, question 2 of the protocol patient survey) with patient report of financial difficulty (as measured by item #28 of the EORTC QLQ-C30). Financial difficulty will be modeled as a latent class predictor within a multinomial logistic regression in addition to the original LCA measurement model. Item #28 on the EORTC QLQ-C30 is measured as "Not at all/A little/Quite a bit/Very much", converted to 0, 1, 2 and 3 respectively for the purposes of analysis. Part 1, question 2 of the protocol patient survey asks the participant if they or anyone in their family have medical bills that they are unable to pay at all.
Proportion of patients who report receiving financial support in the past 12 months | Up to 8 weeks
  The proportion of patients who report receiving financial support (patient survey part 2 question 3 [yes/no]) in the past 12 months will be described using summary statistics.
To describe the association of patient report of receiving financial support with receiving treatment at practices offering patients financial guidance through navigators or social workers, and with socioeconomic status. | Up to 8 weeks
  Logistic regression with receipt of financial support in the past 12 months (patient survey part 2 question 3 [yes/no]) as the dependent variable will be used to test the hypothesis that individuals with multiple myeloma (MM) or chronic lymphocytic leukemia (CLL) will be more likely to report receipt of financial support if they are treated at practices reporting that they offer patients financial guidance through navigators or social workers compared to those treated at practices without these resources. The model will control for disease/treatment characteristics and indicators of patient socioeconomic status.
Patient concerns regarding treatment and costs assessed using aggregate scores of the Valuing Dimensions of the Patient Experience Questionnaire | Up to 8 weeks
  Aggregate scores of the Valuing Dimensions of the Patient Experience Questionnaire measuring patient concerns regarding treatment and costs of care (part 1, questions 22-36 of the protocol patient survey) will be analyzed descriptively. These questions are all assessed as "Very worried", "Somewhat worried" and "Not worried" will be scored as 2, 1 and 0 respectively and aggregated using standard practices.
To describe the association of patient concerns regarding treatment and costs of care with patient socio-demographics, disease characteristics, and practice characteristics. | Up to 8 weeks
  Aggregate scores of the Valuing Dimensions of the Patient Experience Questionnaire measuring patient concerns regarding treatment and costs of care (part 1, questions 22-36 of the protocol patient survey) will be stratified by demographics (e.g. gender, race/ethnicity), socioeconomic characteristics (e.g. education, income), disease characteristics (e.g. MM, CLL), and practice-specific factors (e.g. presence of a social worker/patient navigator). These questions are all assessed as "Very worried", "Somewhat worried" and "Not worried" will be scored as 2, 1 and 0 respectively and aggregated using standard practices. Differences in the aggregate scores between groups will be tested using t-tests. Adjustment for multiple comparisons will not be conducted, which is consistent with social science and/or preference based research.
Association of financial difficulties in past 12 months assessed with EORTC QLQ-C30 and patient health/well-being assessed using Patient-Reported Outcomes Measurement Information System (PROMIS)-10, EuroQol EQ-5D-5L, Brief Appraisal Inventory (BAI) | Up to 8 weeks
  Aggregate scores of the PROMIS-10, EQ-5D-5L and the BAI will be utilized as covariates in a logistic regression model to assess if there is any association with them and the outcome of patient-reported financial difficulty (item #28 of the EORTC QLQ-C30). The PROMIS-10 is a 10-item instrument scored on a scale from 0 - 50 (higher scores = improved QOL). The EQ-5D-5L is a 5-item instrument (5 point scales scored 1-5, where higher scores = worse QOL) and the EQ Visual Analogue scale to score the patient's self-rated health on a scale from 0-100, where higher scores = better QOL. The BAI is a 23-item questionnaire asking patients to rate how often they thought about a variety of topics (Always, Often, Sometimes, Rarely, Never, Not Applicable and Refused to answer). Questions are scored on a scale from 1-5 (Not Applicable and Refused to answer are 88 and 99, respectively, and excluded from scoring), and the questionnaire is scored using standard scoring algorithms.

CONTACTS AND LOCATIONS:
Overall Officials: Rena M. Conti, PhD, Study Chair — Boston University Questrom School of Business
Locations (116):
- United States (116):
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Northside Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Physicians' Clinic of Iowa PC, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - HaysMed University of Kansas Health System, Hays, Kansas
  - Olathe Health Cancer Center, Olathe, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - LSU Health Baton Rouge-North Clinic, Baton Rouge, Louisiana
  - Louisiana Hematology Oncology Associates LLC, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Our Lady of the Lake Physicians Group - Medical Oncology, Baton Rouge, Louisiana
  - Northshore Oncology Associates-Covington, Covington, Louisiana
  - Terrebonne General Medical Center, Houma, Louisiana
  - Ochsner Medical Center Kenner, Kenner, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Saint Joseph Mercy Brighton, Brighton, Michigan
  - Saint Joseph Mercy Canton, Canton, Michigan
  - Saint Joseph Mercy Chelsea, Chelsea, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Ascension Saint Joseph Hospital, Tawas City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Sanford Cancer Center Worthington, Worthington, Minnesota
  - Freeman Health System, Joplin, Missouri
  - Truman Medical Centers, Kansas City, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Community Medical Hospital, Missoula, Montana
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Mission Hospital, Asheville, North Carolina
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - Waverly Hematology Oncology, Cary, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Adena Regional Medical Center, Chillicothe, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Kaiser Permanente Northwest, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Prisma Health Cancer Institute - Laurens, Clinton, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Tidelands Georgetown Memorial Hospital, Georgetown, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - MGC Hematology Oncology-Union, Union, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Regional Cancer Center at Indian Path Community Hospital, Kingsport, Tennessee
  - Wellmont Medical Associates-Bristol, Bristol, Virginia
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Marshfield Clinic Stevens Point Center, Stevens Point, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Conti RM, McCue S, Dockter T, Gunn H, Dusetzina S, Bennett A, Rapkin BD, Gracia G, Jazowski SA, Behrens R, Richardson PG, Chow S, Subbiah N, Neuman HB, Chang GJ, Weiss E. Observational survey of financial difficulties among patients with multiple myeloma and chronic lymphocytic leukaemia treated at US community oncology clinics (Alliance A231602CD). BMJ Open. 2025 Jun 3;15(6):e091769. doi: 10.1136/bmjopen-2024-091769. PMID 40461152